CLINICAL TRIAL: NCT00069069
Title: Induction of Mucosal Tolerance to Human E-Selectin for the Secondary Prevention of Stroke
Brief Title: E-Selectin Nasal Instillation to Prevent Secondary Stroke
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 030293; 03-N-0293
Record Dates: First submitted 2006-07-12; First posted 2003-09-15 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-05-09

CONDITIONS: Ischemic Attack, Transient; Transient
Keywords: Stroke; TIA
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke

ARMS (1):
- 1 (Experimental): single center, Phase 1, open label, dose escalation trial assessing safety profile of four doses of intranasal recombinant human E-selectin
  Interventions: Drug: Intransal instillation of E-selectin

INTERVENTIONS:
Drug: Intransal instillation of E-selectin — Intranasal recombinant human E-selectin

SUMMARY:
This study will determine the maximum safe dose of the experimental drug E-selectin that can be given to stroke patients. E-selectin causes white blood cells called lymphocytes to change so that they prevent clots from forming in the vessels that supply blood to the brain. The drug has been shown to be effective in animal models of stroke. This study will look at the safety of using this experimental drug in nasal instillation form in patients who have had a stroke or transient ischemic attack (TIA).

Patients 45 years of age or older who have had a recent stroke or TIA (30 to 120 days before entering the study) due to a clot forming in a vessel that supplies blood to the brain may be eligible for this study. They must be taking at least one medication to prevent clots, such as coumadin, aspirin, ticlopidine, or others. Candidates will be screened with a physical and neurological examination, blood and urine tests, electrocardiogram (EKG), echocardiogram (ultrasound test of the heart), and magnetic resonance imaging (MRI) of the brain.

Participants will be randomly assigned to receive E-selectin at a dose level of 5, 15, or 50 micrograms or a placebo (nasal drops with no active ingredient). They will instill a small, carefully premeasured amount (one dose) of fluid in their nose every other day for 10 days (total of 5 doses). This course of treatment will be repeated two times at 3-week intervals. Patients will be followed at 1 month and 3 months with a neurologic examination and blood and urine tests. They will be contacted by phone, fax, or email in between these two visits.

DETAILED DESCRIPTION:
In the United States, stroke is the third leading cause of death and the leading cause of disability. Despite the use of antithrombotic drugs for the secondary prevention of stroke, 10% of patients who experience a cerebral ischemic event will go on to have a stroke within 90 days (Claiborne Johnston et al. 2003). The development of new treatment strategies for the secondary prevention of stroke is an important issue for modern medicine. There is increasing evidence that inflammation at the sites of endothelial activation plays an important role in the pathogenesis of stroke. Control of molecular inflammation at the sites of endothelial activation can be achieved by induction of mucosal tolerance. The induction of mucosal tolerance with repeated low-dose intranasal administration of antigen causes a shift of immune response from proinflamatory T helper type 1(T(H)1) effects to anti-inflammatory immunmomodulatory regulatory T cell (Treg) or T helper type 2 (T(H)2) effects at the sites of inflammation. E-selectin is an adhesion molecule expressed only on activated endothelium in response to proinflammatory cytokines.

Objective. The goals of the study are: (a) to test whether repeated administration of low-dose intranasal E-selectin is safe and tolerable and (b) to test whether it can induce mucosal tolerance to this compound causing a shift of immune response from TH1 to TH2 type with production of Treg cells.

Study Population. The study population will include 3-50 patients (depending on dose escalation events) plus 0-8 replacement patients (depending on the number of drop outs) with recent (>30 and <120 days) occurrence of any type or location of stroke documented by CT or MRI. The final number of patients will be determined by a dose escalation plan described below that may stop early in the accrual process should adverse events arise. Since patients will be required to make serial visits to the NIH clinical center, a functional recovery score of 0-2 on the modified Rankin Scale (i.e. 0 = no symptoms at all; 2 = slight disability: unable to carry out all previous activities, but able to look after own affairs without assistance) is required for inclusion in this study.

Study Design. This is a single center, Phase 1, open label, dose escalation trial assessing safety profile of four doses of intranasal recombinant human E-selectin.

Outcome Measures. The primary goal of this study is to define the maximum tolerated dose of intranasal instillation of recombinant human E-selection as described I the Study Medications and Drug Administration section. The secondary goal is to determine doses that generate Treg cells or induce immune deviation from TH1 to TH2 type response. The tertiary goals are to determine the presence or absence of antibody to human E-selectin, P- selectin, and L-selectin and the level of endothelial activation markers including von Willebrand factor, soluble E-selectin, VCAM-1, and Thrombomodulin.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Occurrence of any type or location of stroke (acute ischemic or primary hemorrhagic stroke) at least 31 days, but not more than 120 days prior to enrollment confirmed by brain imaging (CT or MRI).
  2. Age equal to or greater than 45 years.
  3. Modified Rankin Score of 0-2 (functionally independent) at the time of study enrollment and determined to be clinically and neurologically stable by the enrolling investigator.

EXCLUSION CRITERIA:

Patients with any of the following conditions will not be eligible for participation in this study:

1. Intracranial or extracranial dissection, Moyamoya disease, vasculitis, radiation-induced vasculopathy, fibromuscular dysplasia, venous thrombosis.
2. Current treatment with Immunosuppressive medication including: prednisone, cyclophosphamide, cyclosporine, methotrexate, azathioprine, mycophenolate mofetil, anti-CD3 moab (Othoclone OKT3), takrolimus (FK506), sirolimus, anti-IL2r moab (simulect, zenapax), etanercept, infliximab, lenercept, thymoglobulin; thalidomide.
3. Known active autoimmune diseases (RA, LE, MS, Myasthenia Gravis, etc.).
4. Active cancer or lymphoproliferative diseases. (except for basal cell carcinoma)
5. Thrombocytopenia (platelets less than 100,000).
6. HIV or other known immunodeficiencies.
7. Recent major surgery performed within one month of study enrollment.
8. Active systemic infections, or severe focal or upper respiratory infections (URI).
9. Alcohol or substance abuse.
10. Dementia or psychiatric problems (determined by examination, mini-mental status test) that prevents the patient from providing informed consent or following an outpatient program reliably.
11. Pregnancy (urine pregnancy test will be given to women of childbearing potential).
12. Severe rhinopathy or sinusitis.
13. Continuing use of any other over the counter, prescribed or recreational intranasal drug.
14. History of NCI grade 3 epistaxis within 1 month.
15. Exposure to an investigational drug within the 30 days prior to screening for this study.
16. Planned surgery (e.g. carotid or cardiac surgery) or endovascular intervention during the study period until study variables have returned to baseline to prevent attributions of surgical complications to E-selectin tolerization.
17. Patients who are not eligible for or unable to tolerate a brain MRI prior to the start of study drug.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-10-01; Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
To define the MTD for intranasal instillation of recombinant human E-selectin. | One year

SECONDARY OUTCOMES:
Immune deviation from TH1 to TH2 type response with generation of Treg cells. | One year

CONTACTS AND LOCATIONS:
Overall Officials: John M Hallenbeck, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Adams HP Jr, Bendixen BH, Kappelle LJ, Biller J, Love BB, Gordon DL, Marsh EE 3rd. Classification of subtype of acute ischemic stroke. Definitions for use in a multicenter clinical trial. TOAST. Trial of Org 10172 in Acute Stroke Treatment. Stroke. 1993 Jan;24(1):35-41. doi: 10.1161/01.str.24.1.35. PMID 7678184
- [Background] al-Sabbagh A, Nelson PA, Akselband Y, Sobel RA, Weiner HL. Antigen-driven peripheral immune tolerance: suppression of experimental autoimmmune encephalomyelitis and collagen-induced arthritis by aerosol administration of myelin basic protein or type II collagen. Cell Immunol. 1996 Jul 10;171(1):111-9. doi: 10.1006/cimm.1996.0180. PMID 8660845
- [Background] Asai T, Storkus WJ, Whiteside TL. Evaluation of the modified ELISPOT assay for gamma interferon production in cancer patients receiving antitumor vaccines. Clin Diagn Lab Immunol. 2000 Mar;7(2):145-54. doi: 10.1128/CDLI.7.2.145-154.2000. PMID 10702485